CLINICAL TRIAL: NCT04378374
Title: The Effect of Food Formulated With Pulse Flours on Blood Glucose, Satiety and Food Intake
Brief Title: The Effect of Pulse Flours on Blood Glucose, Satiety and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Saint Vincent University (Other)
Responsible Party: Principal Investigator, Bohdan Luhovyy, Associate Professor, Mount Saint Vincent University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2018-201
Record Dates: First submitted 2020-05-02; First posted 2020-05-07 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Blood Glucose; Eating; Appetite; Food
Keywords: Pulses; Flour; Food Intake; Satiety; Blood Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The participants and investigators are blinded and could not distinguish the food formulated with different flours. The taste and flavour in all treatments were similar due to added flavourings.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Baked food made of lentil flour (Experimental): Food prepared with 100% lentil flour
  Interventions: Other: Food-1
- Baked food made of lentil flour and wheat flour (Experimental): Food prepared with a mixture of lentil flour and wheat flour
  Interventions: Other: Food-2
- Baked food made of wheat flour (Experimental): Food prepared with 100% wheat flour
  Interventions: Other: Food-3
- Water (Experimental): Potable water (energy and carbohydrate-free control)
  Interventions: Other: Food-4

INTERVENTIONS:
Other: Food-1 — Baked food made of lentil flour
  Arms: Baked food made of lentil flour
Other: Food-2 — Baked food made of lentil flour and wheat flour
  Arms: Baked food made of lentil flour and wheat flour
Other: Food-3 — Baked food made of wheat flour
  Arms: Baked food made of wheat flour
Other: Food-4 — Potable water (energy and carbohydrate-free control)
  Arms: Water

SUMMARY:
Pulse flours represent a fast-growing segment on the functional food market; however, their health effects are not well understood. The observational studies and acute trials have established the link between frequent consumption of cooked whole pulses (beans, peas, lentils and chickpeas) and healthier body weight and improved blood glucose control. However, it is not clear whether these effects still remain after the processing of pulses into flours. The investigators hypothesized that the baked food products formulated with lentil flour of the same particle size as all-purpose wheat flour may reduce postprandial glycaemia and elicit a stronger suppression of subjective appetite due to its higher content of protein and resistant carbohydrate compared to all-purpose wheat flour. The treatments will be formulated either with lentil flour or with all-purpose wheat flour of similar particle size or with their combination. The objective of the project is to test the effect of foods formulated with lentil flour and/or wheat flour on blood glucose, short-term food intake and subjective appetite.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young male and female adults (19-35 y) with body mass index (BMI) of 20.0-24.9kg/m2

Exclusion Criteria:

* Breakfast skippers
* Smokers (including e-cigarettes) / cannabis consumers
* Those with BMI < 18.5 and > 24.5 kg/m2
* People with chronic diseases
* People with impaired blood glucose control
* People taking medication that may affect central and peripheral mechanisms of food intake regulation, blood glucose control, cognitive performance and sedative medication.
* People with intellectual disabilities (excluded due to their inability to comprehend hedonic and visual analogue scales used in the study).
* People with food allergies or gastrointestinal disorders (e.g., IBS and others).

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | 0-120 minutes
  The concentration of venous blood glucose before and after each treatment consumption
Food Intake | 120 minutes
  The amount of energy (kcal) consumed ad libitum at the test meal (pizza lunch) two hours after each treatment consumption
Subjective Appetite | 0-120 minutes
  The subjective assessment of appetite parameters including desire to eat, fullness, hunger and a prospective food consumption measured with 100 mm Visual Analogue Scales with two opposite statements at each end (e.g., for the hunger scale, 0 mm means not hungry at all, and 100 mm means very hungry).

SECONDARY OUTCOMES:
Physical Comfort | 0-120 minutes
  The subjective assessment of wellness and gastrointestinal symptoms including a feeling of nausea, diarrhea, flatulence, and other parameters measured with 100 mm Visual Analogue Scales with two opposite statements at each end.
Palatability of Food | 5 minutes
  The palatability of the treatments will be measured immediately after consumption with a 100 mm Visual Analogue Scale with two opposite statements at each end or with a 9-point hedonic scale.

CONTACTS AND LOCATIONS:
Overall Officials: Bohdan Luhovyy, PhD, Principal Investigator — Mount Saint Vincent University
Locations (1):
- Mount Saint Vincent University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No